CLINICAL TRIAL: NCT07229339
Title: Phase 2 Trial of Zipalertinib in Patients With Resectable Non-Small Cell Lung Cancer With EGFR Exon 20 Insertion or Uncommon/Compound Mutations
Brief Title: Zipalertinib With Carboplatin and Pemetrexed for the Treatment of Resectable, Stage II-IIIB, Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-1863; NCI-2025-08031 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-11-12; First posted 2025-11-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Lung Non-Squamous Non-Small Cell Carcinoma
MeSH Terms: interventions — Specimen Handling; Carboplatin; Magnetic Resonance Spectroscopy; Pemetrexed; zipalertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Zipalertinib, carboplatin, pemetrexed) (Experimental): NEOADJUVANT: Patients receive zipalertinib PO BID on days 1-21, and carboplatin IV, over 15-60 minutes, and pemetrexed IV, over 10 minutes, on day 1 of each cycle. Cycles repeat every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Within 30 days patients undergo standard of care resection surgery.
  ADJUVANT: Between 4 and 12 weeks after surgery patients receive zipalertinib PO BID on days 1-21 of each cycle. Cycles repeat every 21 days for 13 cycles in the absence of disease progression or unacceptable toxicity.
  Patients undergo PET/CT scan and/or MRI during screening and CT scan and blood and urine sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Pemetrexed; Procedure: Positron Emission Tomography; Drug: Zipalertinib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Pemetrexed — Given IV
  Other Names: MTA; Multitargeted Antifolate; Pemfexy
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Zipalertinib — Given PO
  Other Names: CLN 081; CLN-081; CLN081; EGFR Mutant-specific Inhibitor CLN-081; Mutation-specific EGFR TKI TAS6417; Pan- EGFR Inhibitor CLN-081; Pan-mutation-selective EGFR Inhibitor CLN-081; Pan-mutation-selective EGFR Tyrosine Kinase Inhibitor CLN-081; TAS 6417; TAS-6417; TAS6417

SUMMARY:
This phase II trial tests how well zipalertinib with carboplatin and pemetrexed works in treating stage II-IIIB non small cell lung cancer. that can be removed by surgery (resectable). Zipalertinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Carboplatin is in a class of medications known as platinum-containing compounds. It works in a way similar to the anticancer drug cisplatin, but may be better tolerated than cisplatin. Carboplatin works by killing, stopping or slowing the growth of tumor cells. Pemetrexed is in a class of medications called antifolate antineoplastic agents. It works by stopping cells from using folic acid to make DNA and may kill tumor cells. Giving zipalertinib with carboplatin and pemetrexed may kill more tumor cells in patients with resectable, stage II-IIIB non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the major pathologic response (MPR) rate of neoadjuvant zipalertinib plus carboplatin and pemetrexed chemotherapy at time of surgery in patients with resectable EGFR Ex20ins-mutated or uncommon/compound EGFR-mutated non-squamous non small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of zipalertinib plus chemotherapy as measured by overall response rate (ORR), pathologic complete response (pCR), event-free survival (EFS), and nodal downstaging.

II. To evaluate the safety and tolerability of zipalertinib plus chemotherapy.

EXPLORATORY OBJECTIVE:

I. To assess potential prognostic and predictive biomarkers using circulating tumor deoxyribonucleic acid (DNA) dynamics through next-generation sequencing using the Tempus platform.

OUTLINE:

NEOADJUVANT: Patients receive zipalertinib orally (PO) twice daily (BID) on days 1-21, and carboplatin intravenously (IV), over 15-60 minutes, and pemetrexed IV, over 10 minutes, on day 1 of each cycle. Cycles repeat every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Within 30 days patients undergo standard of care resection surgery.

ADJUVANT: Between 4 and 12 weeks after surgery patients receive zipalertinib PO BID on days 1-21 of each cycle. Cycles repeat every 21 days for 13 cycles in the absence of disease progression or unacceptable toxicity.

Patients undergo positron emission tomography (PET)/computed tomography (CT) scan and/or magnetic resonance imaging (MRI) during screening and CT scan and blood and urine sample collection throughout the study.

After completion of study treatment, patients are followed up at 30 days and every 12 weeks for up to 1 year or until cancer progression or initiation of a new cancer therapy, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent prior to initiation of any study specific activities/procedures
* Male or female ≥ 18 years of age at time of enrollment and willing and able to provide informed consent
* Histologically confirmed non-squamous NSCLC performed within 90 days of enrollment with EGFR Ex20Ins-mutated (addition of 1 or more amino acids) or uncommon/compound EGFR mutations (E709X, G719X, L747X, S758I, and/or L861Q) in tumor tissue or blood; any one of these mutations would qualify if compounded with another EGFR mutation
* Staging positron emission tomography-computed tomography (PET-CT) and brain magnetic resonance imaging (MRI) within 60 days of enrollment demonstrating stage II, IIIA, or IIIB (N2) NSCLC (American Joint Commission for Cancer [AJCC] version [v] 9); mediastinal staging is required by bronchoscopy or mediastinoscopy
* No prior systemic treatment for lung cancer
* Resectable and operable as determined by thoracic surgeon
* At least one measurable lesion according to Response Evaluation Criteira in Solid Tumors (RECIST) 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L
* Platelets ≥ 100 x 10^9/L
* Hemoglobin ≥ 9 g/dL without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
* Glomerular filtration rate (GFR; by Cockroft-Gault or equivalent estimation) ≥ 45 mL/min/1.73 m^2
* Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN) OR direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 ULN with the exception of participants with Gilbert's disease
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x ULN
* International normalized ratio (INR) or prothrombin time (PT), and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless participant is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Able to comply with study requirements
* Female participants may not be pregnant or breastfeeding from initial study visit through a minimum of 1 month after last dose of zipalertinib or 6 months after last dose of chemotherapy, whichever is later
* Adequate pulmonary function as defined by no requirement for oxygen supplementation

Exclusion Criteria:

* Concurrent enrollment in another therapeutic clinical study, unless enrolled only in the follow-up period or an observational study. Use of any antineoplastic therapy must not have been received within 30 days prior to the treatment initiation
* Treatment with live virus, including live-attenuated vaccination, within 30 days prior to the first dose of study treatment. Treatment with inactive vaccines (e.g., non-live or non-replicating agent) and live viral non-replicating vaccines within 3 days prior to first dose of study treatment
* History of active primary immunodeficiency
* Mixed small cell and NSCLC histology
* Stages I, IIIB (N3), IIIC, IVA, and IVB NSCLC, including leptomeningeal carcinomatosis or other central nervous system (CNS) metastases
* History of noninfectious pneumonitis that required the use of systemic corticosteroids, history of interstitial lung disease, treatment-related pneumonitis (any grade), or any evidence of clinically active interstitial lung disease
* Unable to swallow tablets or has any disease or condition that may significantly effect gastrointestinal (GI) absorption of zipalertinib (such as active inflammatory bowel disease, malabsorption syndrome, or prior GI resection)
* History of other malignancy within the past 2 years, with the following exceptions:

  * Malignancy treated with curative intent before enrollment, with no known active disease and felt to be at low risk for recurrence by the treating physician, after discussion with the medical monitor.
  * Adequately treated non-melanomatous skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated cervical carcinoma in situ without evidence of disease.
  * Adequately treated breast ductal carcinoma in situ disease or early stage breast cancer without evidence of disease.
  * Prostatic intraepithelial neoplasia without evidence of prostate cancer, or localized prostate cancer that is adequately treated.
  * Adequately treated urothelial papillary noninvasive carcinoma or carcinoma in situ
* Diagnosis of myelodysplastic syndrome (MDS) requiring active MDS-directed treatment
* History of allogeneic organ transplant
* History of hypersensitivity to carboplatin or pemetrexed or any excipients of zipalertinib
* History of myocardial infarction and/or symptomatic congestive heart failure (New York Heart Association > class II) within 3 months prior to first dose of study treatment
* History of cerebral vascular accident (e.g., stroke or transient ischemic attack) within 3 months prior to first dose of study treatment
* History of uncontrolled seizures
* Human immunodeficiency virus (HIV) infection.

  * Participants with HIV infection on antiviral therapy and undetectable viral load are permitted with a requirement for regular monitoring for reactivation for the duration of treatment on study per local or institutional guidelines
  * HIV screening is not required in the absence of clinical suspicion
* Active hepatitis C infection.

  * Defined as participants with detectable hepatitis C antibody [HCV Ab] and hepatitis C virus [HCV] ribonucleic acid (RNA) viral load above the limit of quantification
  * Participants with presence of HCV antibody (HCV Ab positive) and HCV RNA viral load below the limit of quantification (HCV RNA negative) with or without prior treatment are allowed
* Active hepatitis B infection.

  * Defined as presence of hepatitis B surface antigen [HBsAg-positive] and hepatitis B virus [HBV] DNA viral load above the limit of quantification [HBV DNA positive]
  * Participants with resolved HBV infection defined as absence of HBV surface antigen (HBsAg-negative) and presence of HBV core antibody (anti-HBc positive) followed by an HBV DNA viral load below the limit of quantification (HBV DNA negative) are allowed, with a requirement for regular monitoring for reactivation for the duration of treatment on the study and assessing the need for HBV prophylaxis therapy per local or institutional guidelines.
  * Participants with chronic HBV infection inactive carriers state, defined as presence of HBV surface antigen (HBsAg-positive) and HBV DNA viral load below the limit of quantification (HBV DNA negative) are allowed, with a requirement for regular monitoring for reactivation for the duration of treatment on the study and assessing the need for HBV prophylaxis therapy per local or institutional guidelines
* Any condition (concurrent disease, infection, or comorbidity), in the opinion of the Investigator, that interferes with ability to participate in the study, causes undue risk, or complicates the interpretation of safety data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2027-06-01 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response | At time of surgery
  Defined as ≤10% viable tumor present histologically in the resected tumor specimen after neoadjuvant treatment. A 95% confidence interval for the MPR rate will be calculated using the Clopper-Pearson (exact binomial) method.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years
  Defined as complete response or partial response by Response Evaluation Criteria in Solid Tumors 1.1 criteria. ORR estimate and its associated 95% confidence interval will be calculated. Will compute the proportion of participants achieving complete response (CR) or partial response (PR) and compute 95% confidence intervals using the exact (Clopper-Pearson) confidence intervals.
Pathologic complete response | Up to 2 years
  Defined as no viable tumor present histologically in the resected tumor specimen. Will compute the proportion of participants achieving CR or PR and compute 95% confidence intervals using the exact (Clopper-Pearson) confidence intervals.
Event free survival (EFS) | From cycle 1 day 1 to the earliest date of radiographic progression or recurrence, decision to forgo surgery, or death due to any cause, up to 2 years. Each cycle is 21 days
  Will be analyzed using the Kaplan-Meier method. Median EFS and corresponding 95% confidence intervals will be reported.
Nodal downstaging | From baseline to surgery
  Defined as having N2 or N1 disease prior to the initiation of neoadjuvant treatment with subsequent nodal downstaging to N1 or N0 disease at time or surgery. Will be reported as a percentage of participants who achieve histological downstaging at time of surgery.
Incidence of adverse events | Up to 2 years
  Will be assessed using Common Terminology Criteria for Adverse Events version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Arjan Gower, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States